CLINICAL TRIAL: NCT00892151
Title: Evaluation of GLUCOFACTS® Deluxe Diabetes Management System In a Clinical Setting
Brief Title: Evaluation of GLUCOFACTS® Deluxe Diabetes Management System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTD-2009-01
Record Dates: First submitted 2009-05-01; First posted 2009-05-04 (Estimated); Results first posted 2010-05-18 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intended Users of the Software (Experimental): 10 Healthcare Professionals and 40 persons with diabetes (of which 6 were parents/legal guardians of children with diabetes) using a diabetes data management program.
  Interventions: Device: GLUCOFACTS® Deluxe

INTERVENTIONS:
Device: GLUCOFACTS® Deluxe — Diabetes Data Management Software

SUMMARY:
The purpose of this study is to evaluate a Diabetes management program in the hands of potential users, both health care professionals and lay persons.

DETAILED DESCRIPTION:
Diabetes data management programs upload glucose meter results to computers to provide information at home to lay people with diabetes and their healthcare professionals to manage their diabetes. The study evaluated the subjects' success using the software program with a blood glucose meter to perform specific tasks, such as uploading the meter results, changing program and meter settings, and displaying reports. The study also evaluated the system's ease of use and the acceptability of product labeling.

ELIGIBILITY:
Inclusion Criteria:

Lay users must:

* Be at least 18 years of age (at least 80% must be 55 years or less)
* Have diabetes or be the parent or legal guardian of a child with diabetes who routinely test their blood sugar at home
* Be testing blood sugar at home at least twice daily for at least one month or be the parent or legal guardian of a child who has been testing blood sugar at home at least twice daily for at least one month
* Be able to speak, read, and understand English
* Have experience using PC programs or browsing the internet
* Have utilized diabetes management software at home in the last year (at least 75% of lay users) or be familiar with diabetes management software

HCPs must:

* Have experience using diabetes data management software in the medical office or assist in patients' diabetes disease management using software

Exclusion Criteria:

* Person working for a competitive medical device company
* Person having a cognitive disorder or condition which, in the opinion of the investigator, would put the person at risk or compromise the integrity of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Bailey, MD, Principal Investigator — AMCR Institute
Locations (1):
- AMCR Institute, Escondido, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject was withdrawn for non-compliance. The subject was a parent of a child with diabetes and the 17 year old child was performing the software evaluation instead of the parent. The protocol states that the subjects were to be 18 years and older. The subject was withdrawn from the study and the data was not used in the analysis.
Groups:
- Intended Users of the Software: 10 Healthcare Professionals and 40 persons with diabetes (of which 6 were parents/legal guardians of children with diabetes) used a diabetes data management program.
Period: Overall Study
Arm/Group | Intended Users of the Software
Started | 51
Completed | 50
Not Completed | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Groups:
- Intended Users of the Software: Baseline measures apply to lay persons (n=40) not healthcare professionals in the study.
Arm/Group | Intended Users of the Software
Number analyzed (Participants) | 40
Age, Customized [Median (Full Range); unit: years] — Baseline measures apply to lay persons (n=40) not healthcare professionals in the study. Ages ranged from 18 to 67 years.
  years | 36 [18 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Rated Successful (<=3) at Performing Specific Tasks
Description: Study staff rated participants on their success at perfoming specific tasks. The rating scale was:
  1. = Successful
  2. = Successful after being referred to user instructions
  3. = Successful with verbal assistance or review of part of user instructions (Similar to review of a specific function during a Customer Service call.)
  4. = Unsuccessful (Incorrectly performed part of the testing regimen or required intervention by study staff.)
  5. = Problem encountered with software
Time Frame: 1-2 hours
Population: Note: 2 tasks were performed only by the 10 healthcare professionals. Also, one lay person was withdrawn (leaving 50 participants). The subject was a parent of a child with diabetes;the 17 year old child performed the software evaluation instead of the parent. Data for the subject withdrawn from the study was not used in the analysis.
Measure: Number; unit: participants
Arm/Group | Intended Users of the Software
Number analyzed (Participants) | 50
participants
  Start Glucofacts® Deluxe | 50
  Set up Patient Profile (New User) | 50
  Download CONTOUR meter | 50
  Display the 'standard day' report | 50
  Display the logbook | 50
  Enter a Hemoglobin A1c result to the logbook | 50
  Find A1c result in logbook | 50
  Change Blood sugar (BS) ranges in the software | 50
  Change personal BS ranges in the CONTOUR meter | 50
  Change CONTOUR meter settings | 50
  Download CONTOUR USB meter | 50
  Display the 'Summary' report | 50
  Change CONTOUR USB meter HI and LO settings | 50
  Change CONTOUR USB meter trends length | 50
  Change default BS ranges for patients (HCPs only) | 10
  Find patient in database / view data (HCPs only) | 10

2. Secondary Outcome: Percentage of Participants Who Rated Ease of Performing Specific Tasks As <=3
Description: Subjects rated ease of using the software with respect to specific tasks. The rating scale was:
  1. = Very Simple
  2. = Simple
  3. = Neither Simple nor Difficult
  4. = Difficult
  5. = Very Difficult
Time Frame: 1-2 hours
Population: Note: 2 tasks were performed only by the 10 healthcare professionals. Also, one lay person was withdrawn (leaving 50 participants). The subject was a parent of a child with diabetes; the 17 year old child performed the software evaluation instead of the parent. Data for the subject withdrawn from the study was not used in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Intended Users of the Software
Number analyzed (Participants) | 50
percentage of participants
  Start Glucofacts® Deluxe | 100
  Set up Patient Profile (New User) | 100
  Download CONTOUR meter | 100
  Display the 'standard day' report | 98
  Display the logbook | 100
  Enter a Hemoglobin A1c result to the logbook | 90
  Find A1c result in logbook | 88
  Change Blood sugar (BS) ranges in the software | 92
  Change personal BS ranges in the CONTOUR meter | 98
  Change CONTOUR meter settings | 98
  Download CONTOUR USB meter | 96
  Display the 'Summary' report | 100
  Change CONTOUR USB meter HI and LO settings | 96
  Change CONTOUR USB meter trends length | 98
  Change default BS ranges for patients (HCPs only) | 90
  Find patient in database / view data (HCPs only) | 90

3. Secondary Outcome: Number of Participants Who Rated Clarity and Usefulness of User Instructions as >=3
Description: User instructions included online help, User Guide, and a Quick Reference Guide. Subjects rated their clarity and usefulness and the rating scale was:
  1. = Unacceptable
  2. = Poor
  3. = Good
  4. = Very Good
  5. = Excellent
Time Frame: 1-2 hours
Population: Some subjects had no opinion; the number of subjects that did respond with ratings are identified in parentheses.
Measure: Number; unit: participants
Arm/Group | Intended Users of the Software
Number analyzed (Participants) | 50
participants
  Clarity of instructions in User Guide (n=33) | 33
  Clarity-instruct in Quick Reference Guide (n=35) | 35
  Clarity of the online help (n=35) | 31
  Usefulness of instructions in User Guide (n=30) | 30
  Usefulness-instructions Quick Reference Guide(33) | 33
  Usefulness of the online help (n=31) | 29

ADVERSE EVENTS:
Arm/Group | Intended Users of the Software
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less